CLINICAL TRIAL: NCT00044369
Title: Increased Testicular Cd2+ & Infertility With Varicocele ( a Varicose Vein in the Scrotum)
Brief Title: Role of the Toxic Metal Cadmium in the Mechanism Producing Infertility With a Varicocele
Status: Completed | Type: Observational
Sponsor: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Other Study IDs: 10496-CP-001
Record Dates: First submitted 2002-08-27; First posted 2002-08-28 (Estimated); Last update posted 2006-09-04 (Estimated); Status verified 2006-09

CONDITIONS: Varicocele; Male Infertility; Hypospermatogenesis; Non-Obstructive Azoospermia
Keywords: Varicocele; environmental toxins; male infertility; cadmium
MeSH Terms: conditions — Varicocele; Infertility, Male; Oligospermia

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Varicocele repair

SUMMARY:
Varicose veins in the scrotum (varicocele) are responsible for >20% of male infertility in the US. Varicocele are associated with decreased sperm number and markedly reduced sperm fertilizing ability. Surgical repair or removal of varicocele restores fertility in only 1/3 of cases. The goal of this study is to identify markers that predict the outcome of variocele correction. This would offer considerable health cost savings.

Based on preliminary findings, we will obtain testis biopsies and semen specimens from infertile men with varicocele and prospectively examining the levels of cadmium, a toxic metal, and expression of genes required for normal sperm function. The semen and biopsies will be obtained during clinically dictated procedures. Cadmium and gene expression will be compared with response to varicocele repair (i.e., increased sperm production; pregnancy).

ELIGIBILITY:
* Healthy male with varicocele (grades 2 [palpable] or 3 [visible, palpable]) and no other diagnosed cause for infertility
* Non-smoker
* Actively desiring children but never having initiated a pregnancy
* Female partner having no unresolved fertility issues

Ages: 21 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400
Dates: Start 2000-05; Study Completion 2005-04

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Benoff, PhD, Principal Investigator — North Shore University Hospital
Locations (2):
- United States (2):
  - University of Medicine and Dentistry of NJ, Robert Wood Johnson Medical School at Camden, Camden, New Jersey
  - North Shore University Hospital, Manhasset, New York

REFERENCES:
- [Background] Benoff S, Gilbert BR. Varicocele and male infertility: part I. Preface. Hum Reprod Update. 2001 Jan-Feb;7(1):47-54. doi: 10.1093/humupd/7.1.47. No abstract available. PMID 11212074
- [Background] Benoff S, Hurley IR, Barcia M, Mandel FS, Cooper GW, Hershlag A. A potential role for cadmium in the etiology of varicocele-associated infertility. Fertil Steril. 1997 Feb;67(2):336-47. doi: 10.1016/S0015-0282(97)81921-8. PMID 9022613
- [Background] Benoff S, Cooper GW, Centola GM, Jacob A, Hershlag A, Hurley IR. Metal ions and human sperm mannose receptors. Andrologia. 2000 Sep;32(4-5):317-29. doi: 10.1046/j.1439-0272.2000.00401.x. PMID 11021525
- [Background] Benoff S, Jacob A, Hurley IR. Male infertility and environmental exposure to lead and cadmium. Hum Reprod Update. 2000 Mar-Apr;6(2):107-21. doi: 10.1093/humupd/6.2.107. PMID 10782569